CLINICAL TRIAL: NCT05994989
Title: The Effect of Two Different Tranexamic Acid Dose Regimens on Intraoperative and Postoperative Bleeding in Coronary Artery Bypass Surgery
Brief Title: Two Different Tranexamic Acid Regimens in Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Osman Uzundere, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 5.26.2023/408
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Hemorrhage
Keywords: Tranexamic acid; Coronary artery bypass; Hemorrhage
MeSH Terms: conditions — Postoperative Hemorrhage; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients who have undergone coronary artery bypass surgery and received intravenous tranexamic acid either as a bolus or infusion during the intraoperative period will be included in the study. The cases collected over a period of 6 months will be divided into two groups and compared.
  The first group will consist of patients who receive a 10 mg/kg i.v. bolus of tranexamic acid after anesthesia induction, followed by an 8-hour i.v. tranexamic acid infusion at a dose of 2 mg/kg/hour.
- Group 2: Group 2 will consist of patients who receive three doses of tranexamic acid, 10 mg/kg i.v. bolus after anesthesia induction, in the pump, and after protamine sulfate administration.

SUMMARY:
The primary aim of this study is to observe the effects of two different methods of administering tranexamic acid (i.v. bolus and i.v. infusion) routinely used intraoperatively in cardiovascular surgery, on patients' postoperative bleeding amounts. According to the hypothesis established in this study, it is anticipated that administering tranexamic acid as an i.v. bolus dose followed by an 8-hour continuous infusion will result in a more stable blood level compared to the sole i.v. bolus application, thereby being more effective in influencing postoperative bleeding levels.

The study has been designed as a prospective observational research. The outcomes of two different tranexamic acid protocols applied during cardiovascular surgical procedures will be compared. The first group will consist of patients who receive a 10 mg/kg i.v. bolus of tranexamic acid after anesthesia induction, followed by an 8-hour i.v. tranexamic acid infusion at a dose of 2 mg/kg/hour. Group 2 will consist of patients who receive three doses of tranexamic acid, 10 mg/kg i.v. bolus after anesthesia induction, in the pump, and after protamine sulfate administration.

The cases collected over a period of 14 months will be divided into two groups and compared in terms of intraoperative and postoperative bleeding levels, as well as their need for blood products.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have coronary artery disease requiring coronary artery bypass surgery with cardiopulmonary bypass and received intravenous tranexamic acid either as a bolus or infusion during the intraoperative period will be included in the study.
* Writen consent obtained

Exclusion Criteria:

* Patients operated on for reasons other than coronary artery bypass surgery
* Patients who operated on as emergencies
* Patients who have preoperative liver/renal dysfunction or a history of cerebrovascular events
* Patients under the age of 18
* Patients who have coagulation disorder
* Patients who have a history of allergies
* Pregnancy or lactation
* Disabled in spirit or law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have coronary artery disease requiring coronary artery bypass surgery with cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Postoperative hemorrhage | Postoperative 1st, 6th and 24th hours
  The amount of bleeding within the first 24 hours postoperatively will be compared.

SECONDARY OUTCOMES:
Postoperative hemorrhage | Postoperative first 24 hours
  The amounts of blood and blood products administered within the first 24 hours of postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Yaşargil Education and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guo J, Gao X, Ma Y, Lv H, Hu W, Zhang S, Ji H, Wang G, Shi J. Different dose regimes and administration methods of tranexamic acid in cardiac surgery: a meta-analysis of randomized trials. BMC Anesthesiol. 2019 Jul 15;19(1):129. doi: 10.1186/s12871-019-0772-0. PMID 31307381
- [Background] Zhou ZF, Zhai W, Yu LN, Sun K, Sun LH, Xing XF, Yan M. Comparison of the in-vivo effect of two tranexamic acid doses on fibrinolysis parameters in adults undergoing valvular cardiac surgery with cardiopulmonary bypass - a pilot investigation. BMC Anesthesiol. 2021 Feb 2;21(1):33. doi: 10.1186/s12871-021-01234-8. PMID 33530942
- [Background] Tibi P, McClure RS, Huang J, Baker RA, Fitzgerald D, Mazer CD, Stone M, Chu D, Stammers AH, Dickinson T, Shore-Lesserson L, Ferraris V, Firestone S, Kissoon K, Moffatt-Bruce S. STS/SCA/AmSECT/SABM Update to the Clinical Practice Guidelines on Patient Blood Management. J Extra Corpor Technol. 2021 Jun;53(2):97-124. doi: 10.1182/ject-2100053. No abstract available. PMID 34194077
- [Background] Task Force on Patient Blood Management for Adult Cardiac Surgery of the European Association for Cardio-Thoracic Surgery (EACTS) and the European Association of Cardiothoracic Anaesthesiology (EACTA); Boer C, Meesters MI, Milojevic M, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Pagano D. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):88-120. doi: 10.1053/j.jvca.2017.06.026. Epub 2017 Sep 30. No abstract available. PMID 29029990
- [Background] Madathil T, Balachandran R, Kottayil BP, Sundaram KR, Nair SG. Comparison of efficacy of two different doses of tranexamic acid in prevention of post operative blood loss in patients with congenital cyanotic heart disease undergoing cardiac surgery. Ann Card Anaesth. 2021 Jul-Sep;24(3):339-344. doi: 10.4103/aca.ACA_162_20. PMID 34269265